CLINICAL TRIAL: NCT06912971
Title: Fibromyalgia: The Impact of Self-Knowledge on the Well-Being of People With Fibromyalgia
Brief Title: Fibromyalgia: Impact of Self-Knowledge on Well-Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Ana Isabel Ribeiro Cruz, ANA ISABEL RIBEIRO CRUZ, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-2024
Record Dates: First submitted 2025-03-24; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; self-knowledge; quality of life; Enneagram
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-Knowledge Training Group (Experimental): Participants in this group will undergo a self-knowledge training program based on the Enneagram framework. The program consists of 2 sessions, focusing on self-awareness, emotional regulation, and personal growth.
  Interventions: Behavioral: Self-Knowledge Training Program
- Control Group (No Intervention): Participants in this group will not receive any self-knowledge training during the study period. They will continue with their usual care and will be assessed at the same time points as the intervention group.

INTERVENTIONS:
Behavioral: Self-Knowledge Training Program — The intervention consists of a self-knowledge training program based on the Enneagram framework. Participants attend 7 sessions, focusing on self-awareness, emotional regulation, and personal development. The sessions include theoretical explanations, guided self-reflection exercises, and group discussions to help participants better understand their personality patterns and how these influence their perception of pain and well-being.
  Arms: Self-Knowledge Training Group

SUMMARY:
The goal of this observational study is to evaluate the impact of self-knowledge training on the well-being of individuals with fibromyalgia. The main questions it aims to answer are:

Does self-knowledge training improve participants' perceived quality of life?

Does self-knowledge training influence the way participants manage their fibromyalgia symptoms?

Participants will:

Take part in a structured self-knowledge intervention based on the Enneagram framework.

Complete validated questionnaires before and after the intervention to assess their well-being.

Provide qualitative feedback on their experience with the training.

This study will help understand whether self-awareness strategies can be integrated into non-pharmacological approaches for fibromyalgia management.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fibromyalgia
* Age ≥ 18 years
* Ability to understand and provide informed consent

Exclusion Criteria:

* Cognitive impairment that prevents comprehension of the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-06-18 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Quality of Life (EQ-5D-3L) | Baseline and after completion of the 10-week intervention
  The EQ-5D-3L is a generic instrument for assessing health-related quality of life (HRQoL), comprising five dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each dimension is rated on a 3-level scale (1 = no problems, 2 = moderate problems, 3 = severe problems). The responses generate a health index, where higher scores indicate worse quality of life.
Perceived Quality of Life (EQ-VAS) | Baseline and after completion of the 10-week intervention
  The EQ-VAS is a visual analogue scale measuring self-perceived health status. Participants rate their health on a 0-100 scale (0 = worst imaginable health state, 100 = best imaginable health state). Higher scores indicate better perceived quality of life.
Mental Health - Depression, Anxiety, and Stress (DASS-21) | Baseline and after completion of the 10-week intervention
  The DASS-21 is a 21-item questionnaire assessing symptoms of depression, anxiety, and stress. It includes three subscales (7 items each), rated on a 0-3 scale (0 = does not apply at all, 3 = applies very much or most of the time). Higher scores indicate greater severity of symptoms.

SECONDARY OUTCOMES:
Psychological Flexibility (Psy-Flex Scale) | Baseline and after completion of the 10-week intervention
  The Psy-Flex Scale assesses psychological flexibility, a core construct in Acceptance and Commitment Therapy (ACT). It consists of six items, each representing a fundamental process of psychological flexibility. Responses are rated on a 5-point Likert scale (1 = very rarely, 5 = very frequently). Higher scores indicate greater psychological flexibility.
Self-Reflection and Insight (SRIS Scale) | Baseline and after completion of the 10-week intervention
  The Self-Reflection and Insight Scale (SRIS) evaluates self-reflection and insight through three subscales:
  Engagement in Self-Reflection: Assesses the depth of cognitive and emotional self-examination.
  Need for Self-Reflection: Measures the individual's motivation for self-reflection.
  Insight: Evaluates the individual's level of self-awareness and understanding.
  Each item is rated on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree). Higher scores indicate greater self-reflection and insight.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdade de Medicina da Universidade de Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: Undecided
The decision regarding the sharing of individual participant data has not been finalized. Any future data sharing will be subject to ethical review and compliance with data protection guidelines.